CLINICAL TRIAL: NCT05747443
Title: Multilevel Interventions to Increase Adherence to Lung Cancer Screening
Acronym: Larch
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Fred Hutchinson Cancer Center (Other); Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 220-115.001
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer; Lung Cancer Screening
Keywords: Lung Cancer; Low dose CT (LDCT); Lung Cancer Screening; Stepped Reminders; Educational Video; User centered design; Stakeholders; Evaluation; Qualitative; Patient Partners; Adherence
MeSH Terms: conditions — Lung Neoplasms | interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patient Video only (Experimental): About 3 weeks after the index LDCT, the study Medical Assistant (MA) will deliver a link to the Patient Voices Video, an educational video about lung cancer screening.
  Interventions: Other: Patient Education
- Stepped Reminders only (Experimental): Prior to patient's next LDCT scan is due, MA begins Stepped Reminders intervention:
  MA pends LDCT orders to PCP to sign. MA sends reminders to patient when order is placed and follows up by phone if patient has not scheduled LDCT.
  Interventions: Other: Stepped Reminders
- Patient Video and Stepped Reminders (Experimental): See above. Those assigned to the Patient Video and Stepped Reminders will receive both interventions, as described above.
  Interventions: Other: Stepped Reminders; Other: Patient Education
- Usual Care (No Intervention): Those assigned to the the Usual Care arm will continue to receive usual lung cancer screening care.

INTERVENTIONS:
Other: Stepped Reminders — Stepped Reminders, which directly reminds providers to order the next LDCT scan and then reminds patients they are due and prompts them to schedule LDCT with Radiology.
  Arms: Patient Video and Stepped Reminders; Stepped Reminders only
Other: Patient Education — The Patient Voices Video is an educational video about lung cancer screening.
  Arms: Patient Video and Stepped Reminders; Patient Video only

SUMMARY:
Screening for lung cancer has the potential for a profound public health benefit. Repeat annual screening is necessary for early detection of lung cancer. The investigators will test two interventions which include patient education and reminders to improve adherence to lung cancer screening.

DETAILED DESCRIPTION:
Screening for lung cancer has the potential for a profound public health benefit.

Successful population-based screening requires continuous monitoring to adherence repeat screening in high risk adults to achieve similar results. Repeat annual screening is necessary for early detection of lung cancer. Baseline or first LDCT scans detect prevalent lung cancer, when subsequent screening detects new nodules. However, adherence to screening is low, ranging at 28-38% from centers nationally.

The investigators developed two novel, patient-centered interventions to address patient education and offering reminders for on-time screening. To address these goals, the specific aims are to: 1) Compare effectiveness of two multilevel interventions relative to usual care in improving (a) rates of adherence to lung cancer screening, (b) patient-centered outcomes; and (c) clinic outcomes; and 2) Determine the patient-, clinician-, and system-level factors that influence changes in adherence to inform lung cancer screening programs.

ELIGIBILITY:
Inclusion Criteria:

* KPWA members
* Aged 50-78 years
* Have a negative screening LDCT scan
* Speak English or Spanish
* Meet US Preventive Services Task Force guidelines

Exclusion Criteria:

* Patients who were previously diagnosed with lung cancer,
* Patients who have a positive scan,
* Patients who have an indicator for interpreter services, except for Spanish

Ages: 50 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1837 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2025-07-05 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of repeat annual lung cancer screening | 9-15 months after index LDCT
  Electronic health records will be searched for screening low dose CT (LDCT).

SECONDARY OUTCOMES:
Knowledge of lung cancer screening | 8 weeks after index LDCT
  Knowledge of lung cancer screening eligibility, time to return and cost on patient reported outcomes survey.
Attitudes and beliefs | 8 weeks after index LDCT
  The Lung Cancer Screening Health Belief Scale measures self-efficacy for lung cancer screening. The self-efficacy for lung cancer screening scale ranges from 9-36, with higher scores indicating lower self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Wernli, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vasavada A, Palazzo L, Luce C, Sanchez M, Triplette M, Ralston JD, Carter-Bawa L, Green BB, Gao H, Li CI, Anderson ML, Su YR, Rogers K, Wernli KJ. "It's coming whether we want it to or not": A qualitative exploration of older adults' comfort with and perceptions of technology and digital health. Res Sq [Preprint]. 2025 Nov 19:rs.3.rs-8001649. doi: 10.21203/rs.3.rs-8001649/v1. PMID 41333381
- [Derived] Wernli KJ, Anderson ML, Palazzo L, Luce C, Bezman N, Chin M, Gao H, Ralston JD, Rogers K, Su YR, Triplette M, Carter-Bawa L, Vasavada A, Jordan M, West M, Boler S, Green BB. Effectiveness of Health Communication Intervention to Improve Knowledge on Timeliness to Return for Annual Lung Cancer Screening: The Larch Trial. Chest. 2025 Sep 10:S0012-3692(25)05173-6. doi: 10.1016/j.chest.2025.07.4111. Online ahead of print. PMID 40939933
- [Derived] Luce C, Palazzo L, Anderson ML, Carter-Bawa L, Gao H, Green BB, Ralston JD, Rogers K, Su YR, Tuzzio L, Triplette M, Wernli KJ. A pragmatic randomized clinical trial of multilevel interventions to improve adherence to lung cancer screening (The Larch Study): Study protocol. Contemp Clin Trials. 2024 May;140:107495. doi: 10.1016/j.cct.2024.107495. Epub 2024 Mar 11. PMID 38467273